CLINICAL TRIAL: NCT01467245
Title: Hypercapnia During Thoracoscopy or Open Surgery for Repair of Oesophageal Atresia With Tracheo-oesophageal Fistula or Congenital Diaphragmatic Hernia in Neonates: Pilot Randomised Controlled Trial
Brief Title: Open or Keyhole Surgery Through the Chest for Newborn Babies: Effect on Blood Gases
Acronym: CO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09SG04
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Esophageal Atresia With Tracheo-esophageal Fistula; Congenital Diaphragmatic Hernia
Keywords: Thoracoscopy; congenital diaphragmatic hernia; oesophageal atresia; hypercapnia; acidosis; cerebral oxygenation; neonates
MeSH Terms: conditions — Esophageal atresia with or without tracheoesophageal fistula; Hernias, Diaphragmatic, Congenital; Esophageal Atresia; Hypercapnia; Acidosis | interventions — Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypercapnia during thoracoscopy (Experimental): keyhole surgery through the chest for repair of oesophageal atresia with tracheo-oesophageal fistula or congenital diaphragmatic hernia in neonates
  Interventions: Procedure: Hypercapnia during thoracoscopy
- Open surgery (Experimental): open surgery for repair of oesophageal atresia with tracheo-oesophageal fistula or congenital diaphragmatic hernia in neonates
  Interventions: Procedure: Open surgery

INTERVENTIONS:
Procedure: Hypercapnia during thoracoscopy — keyhole surgery through the chest for repair of oesophageal atresia with tracheo-oesophageal fistula or congenital diaphragmatic hernia in neonates
  Arms: Hypercapnia during thoracoscopy
Procedure: Open surgery — open surgery for repair of oesophageal atresia with tracheo-oesophageal fistula or congenital diaphragmatic hernia in neonates
  Arms: Open surgery

SUMMARY:
This is a pilot randomised controlled trial comparing open versus thoracoscopic surgery for repair of oesophageal atresia with tracheo-oesophageal fistula or congenital diaphragmatic hernia in neonates. Thoracoscopic surgery involves insufflation of carbon dioxide into the thoracic cavity and may therefore cause hypercapnia and acidosis.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with diagnosis of oesophageal atresia with tracheo-oesophageal fistula or congenital diaphragmatic hernia

  ->1.6 Kg
* Conventional ventilation (no high frequency ventilation or iNO) for at least 24 hours.
* FiO2 <0.4
* No requirement for inotropes for at least 24 hours

Exclusion Criteria:

* Late diagnosis (after 1 month of age)
* Major congenital heart defects or pulmonary hypertension
* Bilateral grade IV intraventricular haemorrhage
* Previous ECMO
* FiO2 ≥ 0.4

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Arterial blood carbon dioxide measurement | Intra-operative
  Arterial blood carbon dioxide will be measured during operation as standard of practice by obtaining the blood samples

SECONDARY OUTCOMES:
oxygenation of the brain | Intra-operative and 24 hours post-operatively
  oxygenation of the brain will be measured by a non-invasive technique, near infra-red spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Agostino Pierro, Prof, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Yang EY, Allmendinger N, Johnson SM, Chen C, Wilson JM, Fishman SJ. Neonatal thoracoscopic repair of congenital diaphragmatic hernia: selection criteria for successful outcome. J Pediatr Surg. 2005 Sep;40(9):1369-75. doi: 10.1016/j.jpedsurg.2005.05.036. PMID 16150335
- [Background] Holcomb GW 3rd, Rothenberg SS, Bax KM, Martinez-Ferro M, Albanese CT, Ostlie DJ, van Der Zee DC, Yeung CK. Thoracoscopic repair of esophageal atresia and tracheoesophageal fistula: a multi-institutional analysis. Ann Surg. 2005 Sep;242(3):422-8; discussion 428-30. doi: 10.1097/01.sla.0000179649.15576.db. PMID 16135928
- [Background] Krosnar S, Baxter A. Thoracoscopic repair of esophageal atresia with tracheoesophageal fistula: anesthetic and intensive care management of a series of eight neonates. Paediatr Anaesth. 2005 Jul;15(7):541-6. doi: 10.1111/j.1460-9592.2005.01594.x. PMID 15960636
- [Result] Bishay M, Giacomello L, Retrosi G, Thyoka M, Garriboli M, Brierley J, Harding L, Scuplak S, Cross KM, Curry JI, Kiely EM, De Coppi P, Eaton S, Pierro A. Hypercapnia and acidosis during open and thoracoscopic repair of congenital diaphragmatic hernia and esophageal atresia: results of a pilot randomized controlled trial. Ann Surg. 2013 Dec;258(6):895-900. doi: 10.1097/SLA.0b013e31828fab55. PMID 23604057